CLINICAL TRIAL: NCT03368443
Title: Multiple Practice Contexts to Reduce Context-dependent Learning for Gait Training in People With Parkinson's Disease
Brief Title: Multiple Practice Contexts to Reduce Context-dependent Learning in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201612139RIND
Record Dates: First submitted 2017-12-03; First posted 2017-12-11 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; context-dependent learning; transcranial magnetic stimulation; cognitive function
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-room group (Active Comparator): The participants assigned to the Single-room group will receive treadmill training and overground gait training in one room (Room A) throughout the training sessions.
  Interventions: Behavioral: treadmill training and overground gait training
- Two-room group (Experimental): The participants in the Two-room group will receive treadmill training and overground gait training in 2 rooms (Room A and B) in an alternating order.
  Interventions: Behavioral: treadmill training and overground gait training

INTERVENTIONS:
Behavioral: treadmill training and overground gait training — The participants will be randomized into two different groups, and they will receive treadmill and overground gait training in one or two rooms.

SUMMARY:
Context-dependent learning (CDL) is a phenomenon that an individual demonstrates superior motor performance in the environmental context in which a task was originally learned and practiced, while the performance may decrease if carried out in a novel context. It has often been observed that after individuals with Parkinson's disease (PD) learned how to walk in a clinical setting, they appear to have difficulty generalizing the learned walking ability back to their home or community. To date, no effective intervention approaches have been designed to resolve this CDL for people with PD. One approach that could potentially reduce CDL is to practice a motor task in multiple contexts. Learning a task in multiple contexts would make the participants less likely to rely on the inconsistent ambient contextual information, and could facilitate the generation of stronger motor program and schema. No studies to date have investigated the effects of multiple practice contexts on reducing CDL in people with PD. It is also not clear the characteristics of the participants who would benefit from this type of intervention.

This study aims to investigate the effects of gait training in multiple practice contexts on CDL in individuals with PD. Additionally, this study aims to identify the characteristics of the participants who benefit from the intervention.

Sixty-four participants diagnosed with idiopathic PD will be recruited and randomized into 2 groups: Single-room and Two-room groups. The participants will receive 45 minutes of treadmill training and 15 minutes of over-ground gait training for 12 sessions. Throughout the training sessions, the Single-room group will practice walking in the same room, while the Two-room group will receive gait training in 2 distinct rooms. All participants will be assessed by a blinded evaluator before, immediately after, and 4 weeks after the intervention. The participants will undergo a series of cognitive, motor behavior, and neurophysiological examinations.

Group × time repeated measures analysis of variance (ANOVA) and the partial eta square (η2) will be calculated to determine the intervention effects on the outcome measures. Multiple linear regression analyses will be performed to determine the demographic, cognitive and motor behavior, and neurophysiological characteristics of participants who benefit from the proposed interventions.

DETAILED DESCRIPTION:
Background: Recent evidence suggested that individuals with Parkinson's disease (PD) demonstrated greater context-dependency during motor learning than age-matched non-disabled adults. Context-dependent learning (CDL) is a phenomenon that an individual demonstrates superior motor performance in the environmental context in which a task was originally learned and practiced, while the performance may decrease if carried out in a novel context. It has often been observed that after individuals with PD learned how to walk in a clinical setting, they appear to have difficulty generalizing the learned walking ability back to their home or community. To date, no effective intervention approaches have been designed to resolve this CDL for people with PD.

One approach that could potentially reduce CDL is to practice a motor task in multiple contexts. Based on the research conducted with healthy young adults, learning a task in multiple contexts would make the participants less likely to rely on the inconsistent ambient contextual information. Multiple practice contexts could also facilitate the generation of stronger motor program and schema, leading to better transfer performance and less context-dependency. No studies to date have investigated the effects of multiple practice contexts on reducing CDL in people with PD. It is also not clear the characteristics of the participants who would benefit from this type of intervention.

Objectives: This study aims to investigate the effects of gait training in multiple practice contexts on CDL in individuals with PD. Additionally, this study aims to identify the characteristics of the participants who benefit from the intervention.

Methods: A total of 64 participants diagnosed with idiopathic PD will be recruited and randomized into 2 groups: Single-room and Two-room groups. The participants will receive one-on-one therapy including 45 minutes of treadmill training and 15 minutes of over-ground gait training for a total of 12 sessions. Throughout the 12 training sessions, the Single-room group will practice walking in the same room, while the Two-room group will receive gait training in 2 distinct rooms. All participants will be assessed by a blinded evaluator before, immediately after, and 4 weeks after the intervention. The participants will undergo a series of cognitive, motor behavioral, and neurophysiological examinations. Cognitive assessments will include measures of CDL, Montreal Cognitive Assessment, and the Stroop Color-Word test. Motor behavioral measures will include the Unified Parkinson's Disease Rating Scale, five times sit-to-stand test, 10-meter walk test, timed up and go test, the Activities-Specific Balance Confidence Scale, and Parkinson's Disease Questionnaire-39. Neurophysiological outcomes will be examined with transcranial magnetic stimulation to determine the changes in corticomotor excitability associated with the interventions.

Group × time repeated measures analysis of variance (ANOVA) and the partial eta square (η2) will be calculated to determine the intervention effects on the outcome measures. Multiple linear regression analyses will be performed to determine the demographic, cognitive and motor behavior, and neurophysiological characteristics of participants who benefit from the proposed interventions.

ELIGIBILITY:
Inclusion Criteria:

* able to follow instructions to perform the tasks (Mini Mental State Examination ≥ 24)
* able to read and hear properly without or with aids (e.g., eyeglasses or hearing aids)
* can walk independently with or without devices

Exclusion Criteria:

* has other neurological disorders in addition to PD
* has deep brain stimulation or pacemaker implanted in their body
* has a family-history of epilepsy
* has a self-history of seizure
* has unstable medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-12-25 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Context-dependent learning | 45 mins
  To evaluate context-dependent learning, a finger sequence task has been specially designed. The participants will use an enlarged keyboard to complete the designed computer finger sequence task.
10-Meter Walk Test (10-MWT) | 5 mins
  The walking ability of the participants with PD will be assessed with the 10-MWT. The participants will be instructed to walk along a 10-meter walkway in their comfortable and fastest walking speed. Gait parameters including velocity, stride length, cadence, strike angle and lift-off angle will be calculated.
The Timed Up and Go (TUG) Test | 5 mins
  The participants will initially sit on a comfortable chair with hips and knees flexed at 90°. Upon a 'GO' signal, the participants will stand up from the chair, walk for 3 meters, turn around, walk back to the chair, and sit down. The participants will be instructed to complete the task at their preferred/ comfortable speed. Good to excellent test-retest reliability and inter-rater reliability have been established in people with PD.
Activities-Specific Balance Confidence (ABC) Scale | 5 mins
  The Activities-Specific Balance Confidence (ABC) scale will be used to examine an individual's confidence level of not falling when performing activities of daily living. The ABC Scale contains 16 different activities performed indoors and outdoors. The participants will be asked to rate their confidence level (range from 0% to 100% of confidence) of not falling for each item. An average score of the 16 items (range from 0% to 100%) will be calculated to determine the participant's confidence level of not falling when performing the activities of daily living. The internal consistency and test-retest reliability of the ABC scale in patients with PD were excellent.
Corticomotor excitability | 45 mins
  Transcranial magnetic stimulation (TMS) will be used to evaluate corticomotor excitability. Corticomotor excitability outcomes will include resting motor threshold (RMT), motor evoke potential (MEP), cortical silent period (CSP) duration, short-interval intracortical inhibition (SICI), intracortical facilitation (ICF), and long-interval intracortical inhibition (LICI). The RMT could reflect the membrane excitability of the corticospinal neurons and the cortical interneurons. Peak-to-peak MEP amplitude is an indicator of the integrity and excitability of the corticospinal tract. The CSP is a period when EMG activity being suppressed for a few hundred milliseconds after the MEP, and has often been used as an indicator of the inhibitory mechanism occurs within the corticospinal tract. The SICI, ICF, and LICI have been identified to be good indicators of intracortical inhibition and facilitation.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 10 mins
  The MoCA will be used to evaluate general cognitive function of the participants. It evaluates several cognitive functions including attention, set-shifting, short-term memory, verbal fluency, calculation, orientation, digit span, conceptual thinking, and visuospatial processing skills. The total score of MoCA is 30 with a higher score indicating better cognitive function. The MoCA has good to excellent psychometric properties
The Stroop Color-Word test | 5 mins
  The Stroop Color-Word test will be used to evaluate the changes in executive functions in people with PD. The executive functions involved in the Stroop Color-Word test are selective attention, inhibition, and set-shifting. The Stroop Color-Word test comprises the congruent and incongruent testing conditions. The congruent condition is when the color ink of a word is coherent with the written color name, and the incongruent condition is when the color ink differs from the written color name (e.g., the word 'red' written in blue ink). The participants are instructed to read out the ink color of the word, but not the color word name, as accurately and as fast as possible within 45 seconds.
The Unified Parkinson's Disease Rating Scale (UPDRS) | 10 mins
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a well-established and widely used rating tool for the evaluation of disease severity of PD. The UPDRS consists of 4 sections: 1) Mentation, Behavior, and Mood, 2) Activities of daily living (ADL), 3) Motor examination, and 4) Complications of therapy. In this proposed study, we will only evaluate Part 3 of the scale - the motor disturbances of the patients. The section of "motor examination" contains 18 tests with 33 items (some tests contain movement of the left and right extremities and/or trunk), and each item scores from 0 (absent of the symptom) to 4 (marked in the symptom and present most of the time). The total score ranges from 0 to 132 for Part 3 of the UPDRS with a lower score indicates less PD symptoms and a higher score suggests more severe in PD disease. Internal consistency and validity has been established to be excellent for UPDRS.
Five Times Sit-to-Stand (FTSTS) Test | 5 mins
  During the FTSTS test, the participants will be instructed to stand up from a standardized chair and then sit down 5 times as fast as possible. The lesser amount of times that the participants are able to complete the task safely would indicate better strength of the lower extremities. It was found that the test-retest reliability of the FTSTS test was good, and inter-rater reliability was excellent for patients with PD.
Parkinson's Disease Questionnaire-39 (PDQ-39) | 10 mins
  The PDQ-39 is a self-report questionnaire containing 39 items assessing the impact of PD on quality of life. The PDQ-39 covers 8 dimensions: mobility, activities of daily living, emotional well-being, stigma, cognition, communication, and bodily discomfort. The participants are required to answer the questions based on their experiences in the preceding month prior to the interview. The scoring system for each item ranges from 0 (never have difficulty) to 4 (always have difficulty) with lower scores suggesting better quality of life.
New Freezing of Gait Questionnaire (NFOG-Q) | 5 mins
  The NFOG-Q will be used to evaluate the freezing frequency and severity of the patients with PD. It composes of 3 parts; in the first part, a video clip will be shown to the participants with PD and help to classify whether an individual is a freezer or non-freezer. The second and third part of the questionnaire is designed for freezers only. PartⅡassesses the severity of FoG according to the frequency and duration of the freezing episodes, while PartⅢevaluates the impact of freezing on daily activities, such as walking. The reliability and internal consistency of the NFOG-Q have been well-established for patients with PD.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Yun Lee, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan

REFERENCES:
- [Derived] Lee YY, Tai CH, Fisher BE. Training in Varying Environmental Contexts Facilitates Transfer of Improved Gait Performance to New Contexts for Individuals With Parkinson Disease: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 Oct;103(10):1917-1923. doi: 10.1016/j.apmr.2022.06.010. Epub 2022 Jul 8. PMID 35810822